CLINICAL TRIAL: NCT01192815
Title: A Phase II Study of Erlotinib and Radiation Therapy in Patients With Locally Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: Erlotinib Hydrochloride and Radiation Therapy in Stage III-IV Squamous Cell Cancer of the Head and Neck
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2309; NCI-2010-01885 (Other: NCI/CTRP)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Squamous Cell Carcinoma of the Oropharynx; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Squamous Cell Carcinoma of the Oropharynx; Stage IV Verrucous Carcinoma of the Larynx; Stage IV Verrucous Carcinoma of the Oral Cavity
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride; Radiotherapy, Intensity-Modulated; Pharmacogenomic Testing; Gene Expression Profiling; Radiotherapy, Conformal; Biopsy; Enzyme-Linked Immunosorbent Assay; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive erlotinib hydrochloride orally or via gastrostomy tube once daily in weeks 1-9 and then for 2 years following completion of radiation therapy. Beginning on day 1 of week 2, patients undergo radiation therapy once daily, 5 times a week, for 5-7 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Radiation: intensity-modulated radiation therapy; Other: pharmacogenomic studies; Other: gene expression analysis; Radiation: 3-dimensional conformal radiation therapy; Other: biopsy; Other: pharmacological study; Other: laboratory biomarker analysis; Other: questionnaire administration; Other: enzyme-linked immunosorbent assay; Other: polymorphism analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally or via gastronomy tube
  Other Names: CP-358,774; erlotinib; OSI-774; Tarceva
Radiation: intensity-modulated radiation therapy — IMRT will be given in 35 fractions over 7 weeks. The primary tumor and involved nodes (PTV70) will receive 2 Gy per fractions, intermediate-risk areas (PTV63) will receive 1.8 Gy per fractions, and subclinical disease sites (PTV56) will receive 1.6 Gy perfraction. The total doses will thus be 70 Gy, 63 Gy and 56 Gy, respectively.
  Other Names: IMRT
Other: pharmacogenomic studies — Optional correlative studies
  Other Names: Pharmacogenomic Study
Other: gene expression analysis — Correlative studies
Radiation: 3-dimensional conformal radiation therapy — The initial target volume encompassing the gross and subclinical disease sites will receive 2.0 Gy per fraction, five fractions a week to 54 Gy in 27 fractions in 5.4 weeks. The boost volume covering gross tumor and clinically/radiologically involved nodes will receive boost irradiation for additional 16 Gy at 2.0 Gy. The primary tumor and clinically/radiologically-involved nodes will thus receive 70 Gy in 35 fractions over 7 weeks, and uninvolved upper neck nodes will receive an elective dose of 54 Gy in 5.4 weeks.
  The uninvolved lower neck nodes will receive 2.0 Gy per fraction at 3-cm depth to a total dose of 50 Gy in 25 fractions in 5.0 weeks through a matching AP or AP/PA lower neck field.
  Other Names: 3D-CRT; conformal radiation therapy
Other: biopsy — Optional correlative studies
  Other Names: biopsies
Other: pharmacological study — Optional correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Optional correlative studies
Other: questionnaire administration — Optional ancillary studies
Other: enzyme-linked immunosorbent assay — Optional correlative studies
  Other Names: ELISA
Other: polymorphism analysis — Optional correlative studies

SUMMARY:
RATIONALE: Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Erlotinib hydrochloride may also make tumor cells more sensitive to radiation therapy. Radiation therapy uses high-energy x- rays and other types of radiation to kill tumor cells. Giving erlotinib hydrochloride together with radiation therapy may be an effective treatment for patients with head and neck cancer.PURPOSE: This phase II trial is studying how well giving erlotinib hydrochloride together with radiation therapy works in treating patients with stage III-IV squamous cell cancer of the head and neck.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:I. To determine the time to progression of the combination of the EGFR inhibitor erlotinib and radiation therapy. SECONDARY OBJECTIVES:I. To determine objective response rate, locoregional control rate, duration of response, patterns of failure, overall survival, toxicities and quality of life outcomes of the combination of erlotinib and concurrent radiation therapy.II. To determine the pharmacokinetic profile of erlotinib. Additional analyses of the pharmacokinetic data on patients receiving daily erlotinib treatment via their feeding tube will be conducted. III. To determine the effect of treatment and dose of treatment on biologic correlates in tumor tissue and/or surrounding mucosa, EGFR expression and phosphorylation status, serum markers of angiogenic activity VEGF, sVEGFR-2, sKIT, ICAM, PDGF, fluorescence in situ hybridization (FISH) for ERBB2 for gene amplification, DNA-sequencing of EGFR and ERBB2 genes from DNA extracted from pretreatment biopsy material for mutation screening, gene expression profiling on pre-treatment biopsy material to identify predictors of response to treatment, apoptosis (TUNEL assay), Ki67 (nuclear proliferation antigen)IV. To determine the utility of the comprehensive geriatric assessment, in predicting tolerance to treatment in patients >= 65 years included in this trial. OUTLINE: Patients receive erlotinib hydrochloride orally or via gastrostomy tube once daily in weeks 1-9 and then for 2 years following completion of radiation therapy. Beginning on day 1 of week 2, patients undergo radiation therapy once daily, 5 times a week, for 5-7 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.After completion of study treatment, patients are followed up at 6 months, every 3 months for 2 years, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed locally advanced (stage III or IV) squamous cell carcinoma of the head and neck without distant metastatic disease, who are not candidates or have declined definitive surgical resection or for administration of standard chemotherapy during radiation therapy because of any of the following reasons: advanced age (>= 70 years); poor ECOG performance status (2 or 3); significant comorbidities, as reflected by a Charlson comorbidity index score of >= 3; abnormal hematopoietic, hepatic or renal function; patient's decision after applicable standard treatment options have been offered and declined by patient
* No prior chemotherapy, radiation therapy, or investigational antitumor drug
* Measurable disease within 4 weeks prior to registration according to the recommended RECIST response criteria
* Life expectancy of greater than 12 weeks
* Patients must have normal hepatic function or well compensated liver disease as defined by the Child-Pugh classification of severity of liver disease; patients with hepatic impairment (total bilirubin greater than upper limit of normal [ULN] or well-compensated disease [Child-Pugh class A] enrolled in the trial will be closely monitored, especially those with total bilirubin > 3 times ULN; dosage modifications (therapy interruption or discontinuation) may be necessary for severe changes in liver function; patient management will follow the FDA-approved labeling recommendations
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter
* Women of childbearing potential must have a negative pregnancy test; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* All histologies other than squamous cell carcinoma
* Salivary gland paranasal sinus and nasopharyngeal squamous cell carcinoma
* Patients who have had prior chemotherapy or radiotherapy
* Patients with metastatic disease
* Patients with ECOG performance status of 4
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ERLOTINIB
* Patients with history of any other malignancy (except squamous cell or basal cell cancer of the skin or CIS of cervix) are ineligible unless a period of 5 years has elapsed since treatment of the previous cancer and the patient is currently disease-free from the previous cancer
* Patients may not be receiving any other investigational agent
* Pregnant women; breastfeeding should be discontinued

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panayiotis Savvides, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from local medical clinic from January 2011 through May 2012.
Period: Overall Study
Arm/Group | Arm I
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever status is recorded first) until the first date that recurrence or PD is objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started. Disease progression free survival (PFS) is measured from start of treatment to the date of disease progression or protocol-designated outcome, whichever occurs first and censored at the date of last followed for those survivors without disease progression
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Measured via Conventional CT and MRI
Time Frame: 1 year and 10 months following study start
Population: One patient progressed while study was still active, study closed before follow up completed for second participant and therefore was not evaluable.
Measure: Number; unit: months
Arm/Group | Arm I
Number analyzed (Participants) | 1
months | 6

2. Secondary Outcome: Objective Response Rate
Description: Number of patients with complete response, partial response, stable disease, or progressive disease. Assessed via Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Measured via conventional CT and MRI
Time Frame: 1 year and 10 months following study start
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 1
Participants
  Partial response | 1
  Complete response | 0
  Stable disease | 0
  Progressive disease | 0

3. Secondary Outcome: Patterns of Failure
Time Frame: 5 yrs following treatment
Population: Participants did not complete follow-up per protocol as trial was terminated early
Arm/Group | Arm I
Number analyzed (Participants) | 0

4. Secondary Outcome: Toxicities, Number of Persons With Adverse Events
Description: Number of participants who experienced adverse events (AE's) and serious adverse events (SAE's) during the course of the trial according to CTCAE (4.0)
Time Frame: up to 2 yrs after treatment
Population: Participants enrolled in trial and given treatment. See AE section for details.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 2
Participants | 2

5. Secondary Outcome: Quality of Life Assessment as Measured by Functional Assessment of Cancer Therapy (FACT-G) Test
Description: Quality of Life (QOL) measured using the Functional Assessment of Cancer Therapy-General (FACT-G) on a 0-108 scale, with lower scores corresponding to worse overall QOL and higher scores corresponding to better overall QOL.
Time Frame: after treatment at 6 mos
Population: QOL was no collected and analyzed for this study due to study termination.
Arm/Group | Arm I
Number analyzed (Participants) | 0

6. Secondary Outcome: Locoregional Control Rate
Time Frame: 5 yrs following treatment
Population: Due to the low accrual no data collected.
Arm/Group | Arm I
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Pharmacokinetic Data
Description: Determine the pharmacokinetic profile of erlotinib. Additional analyses of the pharmacokinetic data on patients receiving daily erlotinib treatment via their feeding tube will be conducted.
Time Frame: pre-treatment then weekly
Population: Both participants did not complete treatment per protocol and were not evaluable. No data collected.
Arm/Group | Arm I
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Lab Correlates
Description: Determine the effect of treatment and dose of treatment on biologic correlates in tumor tissue and/or surrounding mucosa.
Time Frame: 2 yrs post concurrent chemo-radiation therapy
Population: Both participants did not complete treatment per protocol and were not evaluable. No data collected.
Arm/Group | Arm I
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from start of study over a 1 year time period.
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=2)
Hypoglycemia (Metabolism and nutrition disorders) | 1
Surgical and medical procedures - Other, specify (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=2)
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Lymphocyte count decreased (Investigations) | 2
Weight loss (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Psychiatric disorders) | 2
Agitation (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Mucosal infection (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Dizziness (Nervous system disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study funding unavailable therefore study terminated early. Both patients did not complete treatment per protocol and were not evaluable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes